CLINICAL TRIAL: NCT00003717
Title: A Phase II Trial of Weekly Paclitaxel Plus Oral Estramustine in Patients With Hormone Refractory Prostate Cancer
Brief Title: Paclitaxel Plus Estramustine in Treating Patients With Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Barnabas Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066826; STBARN-IND-53879; NCI-V98-1509
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Paclitaxel

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than once drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel plus estramustine in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate (PSA and/or objective response) and duration of response to weekly paclitaxel plus estramustine in patients with metastatic hormone refractory prostate cancer. II. Determine the effect on quality of life of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 1 hour weekly for 4 weeks. Patients receive oral estramustine the day before, the day of, and the day after paclitaxel administration each week. Courses repeat every 4 weeks in the absence of unacceptable toxicity and disease progression. A quality of life questionnaire is completed before treatment and 2 months after treatment initiation.

PROJECTED ACCRUAL: A total of 17 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic (D1 or D2) hormone refractory adenocarcinoma of the prostate with one of the following: -Bidimensionally measurable disease -Bone only metastases with rising PSA levels -PSA only disease defined as rising PSA levels with prior confirmation of D1 or D2 disease PSA must be greater than 8 if bone only or PSA only disease Hormone failure defined as progression after treatment with orchiectomy, LHRH agonist, DES alone, or any hormonal treatment in combination with antiandrogen therapy

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: No other active malignancies within the past 5 years except nonmelanomatous skin cancer or other in situ cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy No prior estramustine alone or in combination with other chemotherapy No prior taxanes No more than 1 prior chemotherapy regimen Endocrine therapy: Concurrent primary hormonal therapy allowed (LHRH agonist or orchiectomy) At least 4 weeks since prior antiandrogen therapy with at least 2 rises in PSA levels Radiotherapy: At least 4 weeks since prior radiotherapy At least 8 weeks since prior strontium-89 therapy Surgery: See Disease Characteristics

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 1998-10

CONTACTS AND LOCATIONS:
Overall Officials: Stuart P. Leitner, MD, Study Chair — St. Barnabas Medical Center
Locations (2):
- United States (2):
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey